CLINICAL TRIAL: NCT05936632
Title: Preferences of Individuals in the United States With Personal Experience of Cancer for Certainty Versus Access When Evaluating New Cancer Drugs. A Discrete Choice Experiment.
Brief Title: Preferences for Certainty Versus Access When Evaluating New Cancer Drugs. A Discrete Choice Experiment.
Status: Completed | Type: Observational
Sponsor: London School of Economics and Political Science (Other)
Responsible Party: Principal Investigator, Robin Forrest, Principal Investigator, London School of Economics and Political Science
Other Study IDs: 213621
Record Dates: First submitted 2023-06-26; First posted 2023-07-10 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Cancer
Keywords: Discrete Choice Experiment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Discrete Choice Experiment (DCE) — DCE survey experiment

SUMMARY:
To provide timely access to new treatments, some eligible drugs can be approved despite uncertainty surrounding the level of clinical benefit they offer patients.

It is not currently known if (and under which circumstances) people would prefer to wait to access some new drugs in exchange for greater certainty surrounding their clinical benefit.

This study aims to elicit the preferences of people in the US with experience of cancer for wait times and clinical uncertainty of new drugs.

To elicit this information, in a survey format, respondents will be presented with a hypothetical scenario and asked to state their preferences for new treatments, each with different attributes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals previously or currently diagnosed with any type of cancer.
* Individuals with immediate family members previously or currently diagnosed with any type of cancer.

Exclusion Criteria:

* Individuals without previous or current diagnosis with any type of cancer (themselves or immediate family members).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Online survey panel consisting of a US nationally representative sample (age, gender, income, race/ethnicity, US state).
Sampling Method: Non-Probability Sample
Enrollment: 998 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Preferences for treatment attributes and trade-offs between attributes. | Through study completion, an average of 4-8 weeks.
  Preferences for different treatment attributes (including clinical uncertainty and wait time), and trade-offs between these, using a study-specific Discrete Choice Experiment (DCE) Questionnaire. Preferences are measured on relative utility scale (arbitrary units, no min/max). Utility indicates preference e.g., higher values are more preferred (better).

CONTACTS AND LOCATIONS:
Locations (1):
- London School of Economics, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Forrest R, Lagarde M, Aggarwal A, Naci H. Preferences for speed of access versus certainty of the survival benefit of new cancer drugs: a discrete choice experiment. Lancet Oncol. 2024 Dec;25(12):1635-1643. doi: 10.1016/S1470-2045(24)00596-5. Epub 2024 Nov 18. PMID 39571597